CLINICAL TRIAL: NCT00103506
Title: A Randomized Controlled Study of DOXIL/CAELYX (Doxorubicin HCL Liposome Injection) and VELCADE (Bortezomib) or VELCADE Monotherapy for the Treatment of Relapsed Multiple Myeloma
Brief Title: Study of DOXIL/CAELYX (Pegylated Liposomal Doxorubicin) and VELCADE (Bortezomib) or VELCADE Monotherapy for the Treatment of Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004117; DOXILMMY3001 (Other: Janssen Research & Development, LLC); 2004-001842-34 (EudraCT Number)
Record Dates: First submitted 2005-02-09; First posted 2005-02-10 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Doxil; Caelyx; Doxorubicin; Velcade; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Doxorubicin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VELCADE (bortezomib) monotherapy (Active Comparator): Bortezomib (VELCADE) 1.3 milligram per meter square (mg/m^2) by rapid (bolus) i.v. administration given on Days 1, 4, 8, and 11 of each 21-day cycle for up to 8 cycles.
  Interventions: Drug: Bortezomib (VELCADE)
- DOXIL/CAELYX in combination with VELCADE (bortezomib) (Experimental): Bortezomib (VELCADE) 1.3 mg/m^2 by rapid (bolus) i.v. administration given on Days 1, 4, 8, and 11 of each 21-day cycle for up to 8 cycles. Doxorubicin hydrochloride (DOXIL/CAELYX) 30 mg/m2 by i.v. infusion will be given on Day 4 of every 21-day cycle after the administration of bortezomib (VELCADE) for up to 8 cycles.
  Interventions: Drug: Bortezomib (VELCADE); Drug: Doxorubicin hydrochloride (DOXIL/CAELYX)

INTERVENTIONS:
Drug: Bortezomib (VELCADE) — 1.3 mg/m^2 by rapid (bolus) i.v. administration given on Days 1, 4, 8, and 11 of each 21-day cycle for up to 8 cycles.
  Arms: VELCADE (bortezomib) monotherapy
Drug: Bortezomib (VELCADE) — 1.3 mg/m^2 by rapid (bolus) i.v. administration given on Days 1, 4, 8, and 11 of each 21-day cycle for up to 8 cycles..
  Arms: DOXIL/CAELYX in combination with VELCADE (bortezomib)
Drug: Doxorubicin hydrochloride (DOXIL/CAELYX) — mg/m^2 by i.v. infusion will be given on Day 4 of every 21-day cycle after the administration of bortezomib (VELCADE) for up to 8 cycles.
  Arms: DOXIL/CAELYX in combination with VELCADE (bortezomib)

SUMMARY:
The purpose of this study is to evaluate time to progression, overall survival, response rate and safety for the two open-label treatment groups; DOXIL/CAELYX in combination with VELCADE vs. VELCADE monotherapy.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), parallel-group, open-label (all involved people know the identity of the intervention), multicenter study in 18 countries. A total of 646 patients with multiple myeloma whose disease has progressed after an initial response to at least 1 line of prior therapy or was refractory to initial treatment will be enrolled. The primary endpoint is time to progression (the interval between the date of randomization and the date of disease progression); secondary endpoints are overall survival (the interval between the date of randomization and the patient's death from any cause), response rate (the proportion of patients in the evaluable population who achieved a complete or partial response), and safety. Other study endpoints include patient reported outcomes and exploratory pharmacogenics (to identify genetic markers of response). Patients are assessed for efficacy and safety every 3 weeks until disease progression is documented or for up to 42 weeks from the start of the first dose of study drug. Patients, who do not progress after the 42-week period, are assessed every 6 weeks until disease progression is documented. Efficacy evaluations includes: serum protein electrophoresis, 24-hour urine collection for protein electrophoresis, skeletal survey (plain films), bone marrow biopsy and aspirate, clinical or radiologic assessment of plasmacytomas, and serum calcium. Responses and progressions are assessed objectively by a computer algorithm based on the EBMT criteria. Safety evaluations include adverse event reports, changes in clinical laboratory findings, and tests for cardiac function (multiple gated acquisition scan/echocardiogram and electrocardiogram). Group A: VELCADE monotherapy: VELCADE 1.3 milligram per meter square (mg/m^2) to be administered by i.v. bolus on Days 1, 4, 8, and 11 of each 21-day cycle. Group B: DOXIL/VELCADE combination: treated with VELCADE at the same dose and schedule as specified in Group A. DOXIL/CAELYX 30 mg/m^2 by intravenous infusion given on Day 4 of every 21-day cycle following the administration of VELCADE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who have received at least 1 prior therapy and who have either responded and later had progressive disease or have progressed during their first therapy (primary refractory) are eligible for the study
* Patients who may have received prior doxorubicin but not more than a cumulative dose of 240 milligram per meter square (mg/m^2) doxorubicin, DOXIL, or the equivalent amount of another anthracycline (i.e., 1 mg doxorubicin = 1 mg DOXIL/CAELYX = 1.8 mg epirubicin = 0.3 mg mitoxantrone = 0.25 mg idarubicin)
* Must have normal cardiac function, as evidenced by a left LVEF within institutional normal limits.

Exclusion Criteria:

* History of treatment with VELCADE or progressive disease while receiving an anthracycline-containing regimen
* No change in disease status during initial therapy
* No treatment for malignancy within past 5 yrs (other than multiple myeloma) or progressive disease while receiving anthracycline-containing regimen
* Non-secretory disease
* Myocardial infarct within past 6 months
* No major surgery in past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2004-12; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (108):
- United States (28):
  - Alabaster, Alabama
  - Surprise, Arizona
  - Berkeley, California
  - Loma Linda, California
  - Los Angeles, California
  - Sacramento, California
  - Norwalk, Connecticut
  - Stamford, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Stuart, Florida
  - West Palm Beach, Florida
  - Altanta, Georgia
  - Boise, Idaho
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Minneapolis, Minnesota
  - Hackensack, New Jersey
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - North Charleston, South Carolina
  - Nashville, Tennessee
- Argentina (4):
  - Buenos Aires
  - Ciudad de Buenos Aires
  - La Plata
  - Mendoza
- Australia (5):
  - Adelaide
  - Darlinghurst
  - Melbourne
  - Perth
  - Sydney
- Austria (5):
  - Graz
  - Innsbruck
  - Salzburg
  - Vienna
  - Wels
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Mont-Godinne
- Canada (6):
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - N/a N/a
- Czechia (3):
  - Brno
  - Olomouc
  - Praha 2 N/A
- France (9):
  - Angers Cedex 1 N/A
  - Bobigny
  - Créteil
  - Lille Cedex N/A
  - Nantes
  - Pierre-Bénite
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Israel (6):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Netherlands (10):
  - Amersfoort
  - Amsterdam
  - Amsterdam-Zuidoost
  - Delft
  - Groningen
  - Nieuwegein
  - Nijmegen
  - Rotterdam
  - The Hague
  - Utrecht
- Poland (6):
  - Bialystok
  - Gdansk
  - Lodz
  - Lublin
  - Warsaw
  - Wroclaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Russia (8):
  - Arkhangelsk
  - Izhevsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Obninsk
  - Saint Petersburg
  - Yekaterinburg
- Singapore, Singapore
- South Africa (5):
  - Bloemfontein
  - Cape Town
  - Johannesburg
  - Parktown
  - Pretoria Gauteng
- Spain (3):
  - Barcelona
  - Madrid
  - Salamanca
- United Kingdom (2):
  - Bath
  - London

REFERENCES:
- [Derived] Dimopoulos MA, Orlowski RZ, Facon T, Sonneveld P, Anderson KC, Beksac M, Benboubker L, Roddie H, Potamianou A, Couturier C, Feng H, Ataman O, van de Velde H, Richardson PG. Retrospective matched-pairs analysis of bortezomib plus dexamethasone versus bortezomib monotherapy in relapsed multiple myeloma. Haematologica. 2015 Jan;100(1):100-6. doi: 10.3324/haematol.2014.112037. Epub 2014 Sep 26. PMID 25261096
- [Derived] Sonneveld P, Hajek R, Nagler A, Spencer A, Blade J, Robak T, Zhuang SH, Harousseau JL, Orlowski RZ; DOXIL-MMY-3001 Study Investigators. Combined pegylated liposomal doxorubicin and bortezomib is highly effective in patients with recurrent or refractory multiple myeloma who received prior thalidomide/lenalidomide therapy. Cancer. 2008 Apr 1;112(7):1529-37. doi: 10.1002/cncr.23326. PMID 18300257
- [Derived] Orlowski RZ, Nagler A, Sonneveld P, Blade J, Hajek R, Spencer A, San Miguel J, Robak T, Dmoszynska A, Horvath N, Spicka I, Sutherland HJ, Suvorov AN, Zhuang SH, Parekh T, Xiu L, Yuan Z, Rackoff W, Harousseau JL. Randomized phase III study of pegylated liposomal doxorubicin plus bortezomib compared with bortezomib alone in relapsed or refractory multiple myeloma: combination therapy improves time to progression. J Clin Oncol. 2007 Sep 1;25(25):3892-901. doi: 10.1200/JCO.2006.10.5460. Epub 2007 Aug 6. PMID 17679727

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade (Bortezomib) Monotherapy: Velcade (bortezomib) 1.3 milligram/meter per square (mg/m^2) by rapid (bolus) intravenous (IV) administration given on Day 1, 4, 8, and 11 of each 21-day cycle for up to 8 cycles.
- Doxil/Caelyx Plus Velcade (Bortezomib): Velcade (bortezomib) 1.3 mg/m^2 by rapid (bolus) IV administration given on Day 1, 4, 8, and 11 of each 21-day cycle for up to 8 cycles. Doxorubicin hydrochloride (DOXIL/CAELYX) 30 mg/m^2 by IV infusion will be given on Day 4 of every 21-day cycle after the administration of VELCADE (bortezomib) up to 8 cycles.
Period: Overall Study
Arm/Group | Velcade (Bortezomib) Monotherapy | Doxil/Caelyx Plus Velcade (Bortezomib)
Started | 322 | 324
Completed | 0 | 0
Not Completed | 322 | 324
Not completed — Study closed by sponsor | 34 | 37
Not completed — Death | 257 | 253
Not completed — Lost to Follow-up | 13 | 13
Not completed — Withdrawal by Subject | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Velcade (Bortezomib) Monotherapy | Doxil/Caelyx Plus Velcade (Bortezomib) | Total
Number analyzed (Participants) | 322 | 324 | 646
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.56) | 61.4 (9.61) | 61.4 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 135 | 283
  Male | 174 | 189 | 363
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 6 | 9 | 15
  AUSTRALIA | 31 | 31 | 62
  AUSTRIA | 12 | 6 | 18
  BELGIUM-LUXEMBURG | 6 | 14 | 20
  CANADA | 20 | 23 | 43
  CZECH REPUBLIC | 14 | 22 | 36
  FRANCE | 21 | 28 | 49
  GREAT BRITAIN | 8 | 7 | 15
  ISRAEL | 25 | 21 | 46
  ITALY | 17 | 11 | 28
  NETHERLANDS | 29 | 32 | 61
  POLAND | 35 | 17 | 52
  PORTUGAL | 6 | 14 | 20
  RUSSIA | 38 | 34 | 72
  SINGAPORE | 3 | 2 | 5
  SOUTH AFRICA | 13 | 15 | 28
  SPAIN | 20 | 15 | 35
  UNITED STATES OF AMERICA | 18 | 23 | 41

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Median time to progression of disease is assessed according to International Myeloma Working Group (IMWG) criteria or death from any cause. IMWG criteria: increase of >=25% from lowest level in Serum M-component or (the absolute increase must be >=0.5 gram per deciliter [g/dL]); Urine M component or (the absolute increase must be >=200 milligram per 24 hour. Only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels. The absolute increase >10 mg/dL. Bone marrow plasma cell percentage >=10%. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing. Development of hypercalcemia. Participants who died or dropped out due to any reason without progression will be censored with the day of death or drop-out, respectively and who are alive at the end of the study without any progression was censored with the last available date.
Time Frame: Up to 1 year and 4 months (From date of first participant randomization [20 December 2004] up to interim analysis cut-off date [28 April 2006])
Population: Intent-to-treat (ITT) included all the randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade (Bortezomib) Monotherapy | Doxil/Caelyx Plus Velcade (Bortezomib)
Number analyzed (Participants) | 322 | 324
Months | 6.5 [5.6 to 7.1] | 9.3 [8.2 to 11.1]

2. Secondary Outcome: Overall Survival
Description: The OS is defined as the time from the date of first dose of study drug to date of death from any cause. If the participant is alive or the vital status is unknown, the participant will be censored at the date the participant will be last known to be alive.
Time Frame: Up to 9 years and 5 months (From date of first participant randomization [20 December 2004] to cut-off date for final survival analysis (16 May 2014)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Velcade (Bortezomib) Monotherapy | Doxil/Caelyx Plus Velcade (Bortezomib)
Number analyzed (Participants) | 322 | 324
months | 30.8 [25.2 to 36.5] | 33.0 [28.9 to 37.1]

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 1 year and 11 months (From date of first participant randomization [20 December 2004] to cut-off date for safety update (28 November 2006)
Population: Safety population included all the participants who received at least one dose of study drug. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Velcade (Bortezomib) Monotherapy | Doxil/Caelyx Plus Velcade (Bortezomib)
Number analyzed (Participants) | 318 | 318
Participants | 105 | 120

ADVERSE EVENTS:
Description: Safety population included all the participants who received at least one dose of study drug.
Arm/Group | Velcade (Bortezomib) Monotherapy | Doxil/Caelyx Plus Velcade (Bortezomib)
Serious Adverse Events (participants affected / at risk) | 105/318 | 120/318
Other Adverse Events (participants affected / at risk) | 299/318 | 313/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade (Bortezomib) Monotherapy (N=318) | Doxil/Caelyx Plus Velcade (Bortezomib) (N=318)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 9
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 2 | 0
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 2 | 2
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 2
Nodal Arrhythmia (Cardiac disorders) | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Hypercorticoidism (Endocrine disorders) | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Corneal Erosion (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Retinal Vein Thrombosis (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Faecaloma (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 2
Gastroduodenal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus Paralytic (Gastrointestinal disorders) | 1 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 7
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal Prolapse (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 13
Asthenia (General disorders) | 1 | 2
Catheter Related Complication (General disorders) | 1 | 0
Chest Pain (General disorders) | 3 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 3
General Physical Health Deterioration (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 15
Sudden Cardiac Death (General disorders) | 1 | 0
Sudden Death (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis Acute (Infections and infestations) | 2 | 0
Bronchitis Chronic (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 3
Candidiasis (Infections and infestations) | 0 | 1
Catheter Related Infection (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 1
Diarrhoea Infectious (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Genitourinary Tract Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 3 | 5
Herpes Zoster Disseminated (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Klebsiella Sepsis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 3
Meningitis Bacterial (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Opportunistic Infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumococcal Bacteraemia (Infections and infestations) | 0 | 1
Pneumococcal Sepsis (Infections and infestations) | 1 | 2
Pneumocystis JiroveCI Pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 20 | 16
Pneumonia Aspergillus (Infections and infestations) | 1 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 1
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 2 | 3
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic Embolus (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 4
Urinary Tract Infection (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0
Drug Toxicity (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Skeletal Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 3
Blood Glucose Increased (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 0 | 2
Troponin I Increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 6 | 6
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone Lesion (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Lysis Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Autonomic Neuropathy (Nervous system disorders) | 1 | 0
Balance Disorder (Nervous system disorders) | 1 | 0
Cauda Equina Syndrome (Nervous system disorders) | 2 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Coordination Abnormal (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Lumbar Radiculopathy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 2
Paralysis (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1
Polyneuropathy in Malignant Disease (Nervous system disorders) | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 3
Syncope (Nervous system disorders) | 4 | 4
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephritis Interstitial (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 2 | 3
Renal Failure Acute (Renal and urinary disorders) | 5 | 4
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 2 | 0
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epidermal Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Jessner's Lymphocytic Infiltration (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 4
Orthostatic Hypotension (Vascular disorders) | 2 | 2
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade (Bortezomib) Monotherapy (N=318) | Doxil/Caelyx Plus Velcade (Bortezomib) (N=318)
Anaemia (Blood and lymphatic system disorders) | 67 | 80
Leukopenia (Blood and lymphatic system disorders) | 23 | 28
Neutropenia (Blood and lymphatic system disorders) | 71 | 113
Thrombocytopenia (Blood and lymphatic system disorders) | 89 | 104
Conjunctivitis (Eye disorders) | 17 | 24
Abdominal Pain (Gastrointestinal disorders) | 23 | 32
Abdominal Pain Upper (Gastrointestinal disorders) | 13 | 24
Constipation (Gastrointestinal disorders) | 98 | 99
Diarrhoea (Gastrointestinal disorders) | 122 | 142
Dyspepsia (Gastrointestinal disorders) | 13 | 27
Nausea (Gastrointestinal disorders) | 125 | 152
Stomatitis (Gastrointestinal disorders) | 11 | 55
Vomiting (Gastrointestinal disorders) | 67 | 93
Asthenia (General disorders) | 56 | 70
Chills (General disorders) | 18 | 25
Fatigue (General disorders) | 88 | 115
Influenza Like Illness (General disorders) | 13 | 18
Oedema Peripheral (General disorders) | 27 | 32
Pyrexia (General disorders) | 67 | 91
Bronchitis (Infections and infestations) | 14 | 25
Herpes Simplex (Infections and infestations) | 18 | 32
Herpes Zoster (Infections and infestations) | 26 | 30
Nasopharyngitis (Infections and infestations) | 20 | 25
Pneumonia (Infections and infestations) | 9 | 18
Upper Respiratory Tract Infection (Infections and infestations) | 32 | 30
Aspartate Aminotransferase Increased (Investigations) | 11 | 16
Blood Creatinine Increased (Investigations) | 7 | 16
Weight Decreased (Investigations) | 12 | 37
Anorexia (Metabolism and nutrition disorders) | 43 | 58
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 30
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 34
Back Pain (Musculoskeletal and connective tissue disorders) | 37 | 38
Bone Pain (Musculoskeletal and connective tissue disorders) | 25 | 10
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 12 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 10
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 47 | 34
Dizziness (Nervous system disorders) | 27 | 32
Dysgeusia (Nervous system disorders) | 9 | 18
Headache (Nervous system disorders) | 56 | 59
Neuralgia (Nervous system disorders) | 63 | 54
Neuropathy (Nervous system disorders) | 38 | 35
Neuropathy Peripheral (Nervous system disorders) | 46 | 36
Paraesthesia (Nervous system disorders) | 31 | 41
Peripheral Sensory Neuropathy (Nervous system disorders) | 42 | 41
Polyneuropathy (Nervous system disorders) | 27 | 26
Depression (Psychiatric disorders) | 16 | 9
Insomnia (Psychiatric disorders) | 43 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 58
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 28
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 62
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 20
Rash (Skin and subcutaneous tissue disorders) | 29 | 48
Hypertension (Vascular disorders) | 17 | 15

LIMITATIONS AND CAVEATS:
Study stopped in terms of primary endpoint based on its results at planned interim analysis (28 Apr 2006). However, Long-term follow-up for survival continued until 16 May 2014.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.